CLINICAL TRIAL: NCT05677997
Title: Evaluating the Impact of Resource Navigators to Support Long-term Care and Retirement Home Staff During and Beyond COVID-19
Brief Title: Evaluating the Impact of Resource Navigators to Support LTC and RH Staff During and Beyond COVID-19
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 22-026
Record Dates: First submitted 2022-12-09; First posted 2023-01-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-05

CONDITIONS: Wellness; Burnout, Caregiver; Burnout, Professional; COVID-19; Vaccine Refusal
Keywords: Caregiver; Personal support worker; long term care home; mental health
MeSH Terms: conditions — Caregiver Burden; Burnout, Professional; COVID-19; Vaccination Refusal; Psychological Well-Being | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Receiving monthly resources only
- Intervention Group (Experimental): Receiving sessions with a resource navigator 2x a month, and monthly resources.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Sessions to go through goals, problem areas, areas they want to improve.
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to test how well resource navigators help long-term care and retirement home staff access the various health and wellness resources available to them and the effects that this has on their health and wellness overall. The main questions it aims to answer are:

- How does one-on-one support from a resource navigator affect the wellness of long-term care and retirement home staff, including burnout, vaccination status, and COVID-19 infection? Researchers will compare participants in the intervention group (where participants are paired with a resource navigator) and the control group (where participants are not paired with a resource navigator) to see the impact access to a resource navigator has on wellness (primary outcome), burnout, knowledge of, access to and use of wellness resources, knowledge/alignment with provincial public health guidelines related to SARS-CoV-2 vaccine outcomes, SARS-CoV-2 infection, hospitalization, and death (secondary outcomes).

Hypothesis: Researchers anticipate that those in the intervention group (have access to a resource navigator) will report a higher positive change in wellness between baseline and 6 months.

DETAILED DESCRIPTION:
In response to the increased stress and workload of the COVID-19 pandemic response for long term care home (LTCH) and retirement home (RH) staff, the Knowledge Translation Program (KTP) at St. Michaels Hospital launched efforts to support this population. Via in-depth discussions and surveys, >200 personal support workers (PSWs) were canvassed to identify their needs during the pandemic. Four areas of need were identified, which included supports for:

1. Wellness, burnout and mental health
2. Infection Prevention and Control (IPAC)
3. Wraparound resources (e.g., access to food banks, caring for a family member with COVID-19) and
4. Vaccine information

Additionally, using the Theoretical Domains Framework, the KTP identified the following barriers that impact PSWs' and/or other long-term care and retirement home staff's ability to navigate the pandemic [1]:

* lack of knowledge of available resources
* perceptions of identity within the long-term care home context, resource challenges (e.g., lack of occupational health programs), and * impact of social influences on beliefs (e.g., family and peer perceptions of vaccine efficacy and safety).

These barriers were mapped to corresponding implementation strategies via the Behaviour Change Wheel framework to identify education and enablement (e.g., supporting individuals' own self-efficacy) as interventions to mitigate the identified barriers.[1] Utility of these interventions was confirmed by long-term care home staff partners who believed routine check in calls would reduce social isolation and support PSWs and other long-term care staff to find and use available resources to address their needs.[1]

Through funding from the COVID-19 Immunity Task Force (CITF), the Ontario Ministry of Labour Training and Skills Development (MOLTSD) and the Canadian Immunization Research Network (CIRN), the KTP developed educational resources compiled in a single online repository for long-term care home staff on optimizing infection prevention and control (IPAC) [2-5] in long-term care home, promoting wellness and preventing burnout [6, 7] providing 'wraparound' [8 ,9] resource supports to individuals (e.g., access to food banks, resources on self-isolation, caring for a family member with COVID-19), and addressing SARS-CoV-2 vaccine [10-12] myths and questions (via infographics and town halls created in partnership with OPSWA).[13, 14]

However, currently long-term care and retirement home staff access these resources passively and many do not have the capacity or skills to implement the resources effectively.

A navigator is the missing link to putting these resources into practice.

Through this clinical trial, the researchers aim to answer the following research question:

What is the impact of tailored 1:1 support from a resource navigator and educational resources (intervention arm) compared to educational resources only (control arm) on the wellness of long-term care and retirement home staff (primary outcome), burnout, knowledge of, access to and use of wellness resources, SARS-CoV- 2 vaccination status, self-reported SARS-CoV-2 infection and hospitalization (secondary outcomes).

To achieve the study aim, the researchers will:

1. Conduct a trial, which will randomize PSWs and other support service staff to receive 6 months of tailored 1:1 support from a resource navigator and educational resources (intervention arm) versus educational resources only (control arm) to navigate the pandemic.
2. Evaluate the impact of the intervention on PSW's and other support service staff's wellness (primary outcome), burnout, knowledge of, access to and use of wellness resources, alignment of provincial public health guidelines related to SARS-CoV-2 vaccine outcomes, SARS-CoV-2 infection, hospitalization, and death (secondary outcomes).
3. Conduct a process evaluation to assess quality and delivery of the study intervention.

This study will take place in Long-Term Care and Retirement Homes in Ontario. Each month, participants in the intervention arm will receive a PDF package by email from a research staff member, which will include wellness, burnout and mental health resources (e.g., how to use the free, self-referral Centre for Addiction and Mental Health service [6]; tips on reducing/preventing burnout [9]), SARS-CoV-2 vaccine infographics [10], a wraparound [8] resource package, and IPAC [5] tips/guidance. Participants that indicated they would like a print copy of the resources in the pre-screening survey will be provided a copy via mail. Participants will also receive two hours (2, 1-hour sessions) of navigation support sessions from the resource navigator (by phone/zoom) per month for six months (Total 12, 1-hour sessions). While the resource navigator will not directly provide counselling or mental health supports, they will serve as a liaison to link the PSWs and other support service staff (where applicable) to these supports. The resource navigators will hold a degree or diploma in social services/work, psychology or a related field and have at least 2 years of experience in these sectors.

In the control arm, participants will receive the monthly educational resources only.

Both intervention and control arms will complete a baseline survey, exit survey (at 6 months), and interview if selected to participate.

ELIGIBILITY:
Inclusion Criteria:

1. A fulltime or part-time employee aged 18 years and older identified as a Long-Term Care and Retirement Home staff (PSW's and other support service staff in those in nutrition, housekeeping and laundry)
2. Work in an Ontario Long-term care or retirement home;
3. Comfortable speaking and reading English; and
4. Access to and willingness to use email for study communications

Exclusion Criteria:

1. Do not identify as or are not employed as a PSW and other support service staff;
2. Do not work in an Ontario long-term care or retirement home;
3. Uncomfortable speaking or reading English; and
4. Do not have access to or unwillingness to use email for study communications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Change in Wellness | Baseline, and 6 months.
  Participant wellness will be assessed using the Personal Wellbeing Score. Survey includes 5 questions and will be scored on a scale from 0 to 16, where 16 is the worst outcome, or poorest level of wellness. For ONS4 life satisfaction, worthwhile and happiness scores, responses 9-10 are grouped as Very high, 7-8 as High, 5-6 as Medium and 0-4 as Low. For anxiety scores, responses 6-10 are grouped as High, 4-5 as Medium, 2-3 as Low and 0-1 as Very low.

SECONDARY OUTCOMES:
Rate of Change in Level of Burnout | Baseline, and 6 months.
  Burnout will be assessed with the 22-item Maslach Burnout Inventory for Medical Personnel. The questionnaire has three main areas which are to be scored independently: emotional exhaustion, on a scale of 0 to 54, where 54 is the worse outcome (highest level of emotional exhaustion); depersonalization, on a scale of 0 to 30, where 30 is the worst outcome (highest level of depersonalization); and low sense of personal accomplishment, on a scale of 0 to 48, where 0 is the worst outcome (lowest sense of personal accomplishment).
Rate of Changes in knowledge, access to and use of wellness supports, | Baseline, and 6 months.
  There are five individual surveys assessing changes to participants' knowledge, access to, and use of wellness supports.
Rate Changes in number of participants with COVID-19 vaccination, number of participants with COVID infection and hospitalization, over time | Baseline, and 6 months.
  Via participants' Ontario Health Insurance Plan (OHIP) number, we will link to the ICES provincial administrative database to obtain participants' vaccine status, and rates of SARS-CoV-2 infection, hospitalization and death.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michaels Hospital,, Toronto, Ontario, Canada

REFERENCES:
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Rios P, Radhakrishnan A, Thomas SM, Darvesh N, Straus SE, Tricco AC. Preventing respiratory illness in older adults aged 60 years and above living in long-term care. MedRxiv. 2020; 1-25. https://doi.org/10.1101/2020.03.19.20039081
- [Background] Rios P, Radhakrishnan A, Williams C, Ramkissoon N, Pham B, Cormack GV, Grossman MR, Muller MP, Straus SE, Tricco AC. Preventing the transmission of COVID-19 and other coronaviruses in older adults aged 60 years and above living in long-term care: a rapid review. Syst Rev. 2020 Sep 25;9(1):218. doi: 10.1186/s13643-020-01486-4. PMID 32977848
- [Background] IPAC+ Self-Assessment for Long-term Care Facilities (LTCHs) and Retirement Homes (RHs). https://ipac.knowledgetranslation.ca/. Accessed 2021 Feb 18.
- [Background] IPAC+ Resource Library. Regional Geriatric Program of Toronto. https://www.rgptoronto.ca/resources/ipac+/. Updated 2021.
- [Background] Mental Health and COVID-19. Centre for Addiction and Mental Health (CAMH). https://www.camh.ca/en/health-info/mental-health-and-covid-19/information-for-professionals. Published 2020.
- [Background] Mental Health Supports. Wellness HUB Support for Congregate Living Centres. https://wellness-hub.ca/tag/mental-health-supports/. Published 2021.
- [Background] Wraparound Resources Package. Wellness Hub. https://wellness-hub.ca/res/wraparound-resources-package/. Published 2021.
- [Background] Caregiver Resources. The Ontario Caregiver Organization. https://ontariocaregiver.ca/resources-education/caregiver-resources/#caring-for-yourself. Published 2021.
- [Background] What you need to know about getting the COVID-19 vaccine. Wellness Hub. https://wellness-hub.ca/res/what-you-need-to-know-about-getting-the-covid-19-vaccine/. Published 2021.
- [Background] February 2nd, 2021 OPSWA Town Hall #2: COVID vaccine questions answered. Knowledge Translation Program. https://www.youtube.com/watch?v=UCzRgtbHFFQ&t=517s. Published 2021 Mar 31.
- [Background] March 23rd, 2021 OPSWA Town Hall #3: Get you COVID vaccine questions answered. Knowledge Translation Program. https://www.youtube.com/watch?v=hNrNsTXKGT8&t=3s. Published 2021 Mar 26.
- [Background] Knowledge Translation Program. COVID-19 Knowledge Translation. https://knowledgetranslation.net/expertise/covid-19/. Updated 2021.
- [Background] COVID-19 Immunity Task Force. Pan-Canadian studies investigate why COVID-19 has been devastating to long-term care facility residents and staff.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT05677997/Prot_SAP_000.pdf